CLINICAL TRIAL: NCT00277264
Title: Spiriva® Assessment of FEV1 (SAFE). The Effect of Inhaled Tiotropium Bromide (18 Mcg Once Daily) on the Change in FEV1 During Long-term Treatment in Patients With COPD. A One-year Parallel Group, Double-blind, Randomised, Placebo-controlled Study
Brief Title: Spiriva® Assessment of FEV1 (SAFE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.259
Record Dates: First submitted 2006-01-09; First posted 2006-01-16 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: Tiotropium (Spiriva®)

SUMMARY:
The objective of this trial is to evaluate whether the effect of one year (48 weeks) treatment with inhaled tiotropium bromide (Spiriva® - 18 µg once daily) on the change in trough FEV1, compared to placebo in patients with COPD, is affected by smoking status.

DETAILED DESCRIPTION:
This was a multi-centre, randomised, double-blind, placebo-controlled study. The duration of subject participation was 48 weeks. There was an initial screening period of up to 2 weeks. The first screening visit consisted of medical history, clinical assessment, safety laboratory assessments and complete pulmonary function testing. The screening period was followed by a randomised treatment period where patients received tiotropium (Spiriva) or placebo in a ratio of 2:1. During the treatment period there were a total of 5 clinic visits (including randomisation and EOT visit). Each visit included lung function measurements and clinical assessments (SQRQ, COPD Symptom scores, physician's global assessment, COPD exacerbations/hospitalisations, vital signs and rescue medication use) in addition to adverse event reporting. The final visit consisted of a telephone contact 2 weeks after the patient completed their trial medication.

Study Hypothesis:

The primary purpose of this trial was to evaluate whether the effect of inhaled tiotropium (Spiriva®) on the change in trough FEV1, compared to placebo, was affected by smoking status. The primary endpoint was defined as the change in trough FEV1 after 48 weeks of treatment. The primary analysis was performed in a sequential fashion; firstly, the analysis was performed for all patients and if a positive signal was seen in this group, the analysis was then performed for both the smoking and ex-smoking groups separately. Patients were defined as smokers or ex-smokers at the screening visit.

Comparison(s):

Tiotropium (Spiriva®) vs placebo

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Stable airway obstruction
* FEV1 < or equal to 65% of predicted
* Male or female
* Age > or equal to 40 years
* > or equal to 10 pack year smoking history
* History of exacerbations in the past year
* Able to be trained in the proper use of the HandiHaler®

Exclusion Criteria:

* History of asthma
* Allergic rhinitis or atopy
* Unstable use (6 weeks) of OCS (or > 10 mg daily use)
* History of life threatening bronchial obstruction, cystic fibrosis or bronchiectasis
* Patients who had started or stopped an exercise rehabilitation program in the past twelve months
* Thoracotomy with pulmonary resection or lobectomy (LVRS)
* Active tuberculosis
* Use of beta-blockers
* Pregnant, nursing women and women of childbearing potential not using a medically approved means of contraception
* 6 months or less history of myocardial infarction
* Intolerance to anticholinergic containing products, and/or to lactose or any other components of the inhalation capsule delivery system
* History of unstable arrhythmia with a life threatening event or change of related therapy during the past year
* History of cancer, other than treated basal cell carcinoma, within the last 12 months
* Clinically relevant abnormal baseline haematology, blood chemistry or urinalysis
* Patients with narrow angle glaucoma
* Patients with symptomatic benign prostatic hypertrophy
* Patients with bladder neck obstruction
* Patients that planned to be out of the country for 8 weeks or more

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 914
Dates: Start 2002-01; Primary Completion 2004-05 (Actual); Study Completion 2004-05

PRIMARY OUTCOMES:
The primary efficacy endpoint was the change in trough FEV1 after 48 weeks of treatment. | after 48 weeks of treatment

SECONDARY OUTCOMES:
The change from baseline FEV1 at interim visits | at Week 2, 11, 30 and 48
The change from baseline FVC | at Week 2, 11, 30 and 48
The change from baseline FEV6 (at selected sites) | at Week 2, 11, 30 and 48
Incidence, severity and duration of COPD exacerbations | at Week 2, 11, 30, 48 and 50
Incidence and duration of hospitalisations due to COPD exacerbations | at Week 2, 11, 30, 48 and 50
Use of rescue medication (day-time and night-time) during treatment period | week 1 until week 48
Number of short courses of steroids/antibiotics during treatment period | week 1 until week 48
Assessment of COPD symptoms | at Week 2, 11, 30 and 48
Physician's Global Evaluation | baseline and week 48
Quality of life questionnaire (SGRQ) | at week 30 and 48
Adverse events | 27 months
Vital Signs | 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Canada Ltd.
Locations (77):
- Canada (77):
  - Respiratory Research, Room 1742, Calgary, Alberta
  - Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 4A-185, 7007-14 Street SW, Calgary, Alberta
  - Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - Boehringer Ingelheim Investigational Site, Lethbridge, Alberta
  - Boehringer Ingelheim Investigational Site, Medicine Hat, Alberta
  - 301-131 First Ave., Spruce Grove, Alberta
  - Boehringer Ingelheim Investigational Site, Wetaskiwin, Alberta
  - Boehringer Ingelheim Investigational Site, Abbotsford, British Columbia
  - Boehringer Ingelheim Investigational Site, Chilliwack, British Columbia
  - Boehringer Ingelheim Investigational Site, Kelowna, British Columbia
  - Boehringer Ingelheim Investigational Site, Maple Ridge, British Columbia
  - 220 Royal Avenue, New Westminster, British Columbia
  - Penticton Regional Hospital, Penticton, British Columbia
  - Boehringer Ingelheim Investigational Site, Surrey, British Columbia
  - Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - Boehringer Ingelheim Investigational Site, Steinbach, Manitoba
  - 1095 Concordia Avenue, Winnipeg, Manitoba
  - Boehringer Ingelheim Investigational Site, Saint John, New Brunswick
  - Boehringer Ingelheim Investigational Site, Mount Pearl, Newfoundland and Labrador
  - 262 Newfoundland Drive, St. John's, Newfoundland and Labrador
  - 300 Prince Philip Drive, St. John's, Newfoundland and Labrador
  - Boehringer Ingelheim Investigational Site, New Glasgow, Nova Scotia
  - Boehringer Ingelheim Investigational Site, Sydney, Nova Scotia
  - Boehringer Ingelheim Investigational Site, Ajax, Ontario
  - Boehringer Ingelheim Investigational Site, Corunna, Ontario
  - Boehringer Ingelheim Investigational Site, Courtice, Ontario
  - 169 Main Street East, Grimsby, Ontario
  - 237 Barton Street East, Hamilton, Ontario
  - HGH McMaster Clinic, Hamilton, Ontario
  - Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 50 Charlton Avenue East, Hamilton, Ontario
  - Boehringer Ingelheim Investigational Site, Kingston, Ontario
  - Boehringer Ingelheim Investigational Site, Kitchener, Ontario
  - Boehringer Ingelheim Investigational Site, London, Ontario
  - Haemolology Division, London, Ontario
  - St Joseph's Healthcare, London, Ontario
  - Boehringer Ingelheim Investigational Site, Markham, Ontario
  - Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 300-2338 Hurontario Street, Mississauga, Ontario
  - Boehringer Ingelheim Investigational Site, Niagara Falls, Ontario
  - Boehringer Ingelheim Investigational Site, North York, Ontario
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - 1053 Carling Avenue, Ottawa, Ontario
  - Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - Boehringer Ingelheim Investigational Site, Peterborough, Ontario
  - Boehringer Ingelheim Investigational Site, Richmond Hill, Ontario
  - Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - Boehringer Ingelheim Investigational Site, Scarborough Village, Ontario
  - Boehringer Ingelheim Investigational Site, Thunder Bay, Ontario
  - Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 825 Coxwell Avenue, Toronto, Ontario
  - 600 Sherbourne Street, Suite 402, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - 76 Grenville Street, Toronto, Ontario
  - Boehringer Ingelheim Investigational Site, Trenton, Ontario
  - Boehringer Ingelheim Investigational Site, Windsor, Ontario
  - Boehringer Ingelheim Investigational Site, York, Ontario
  - 91 Thomas-Chapais, Boucherville, Quebec
  - 305 rue Saint-Vallier, Chicoutimi, Quebec
  - Boehringer Ingelheim Investigational Site, Gatineau, Quebec
  - 4 rue Robinson, Granby, Quebec
  - Boehringer Ingelheim Investigational Site, Greenfield Park, Quebec
  - Boehringer Ingelheim Investigational Site, La Malbaie, Quebec
  - Boehringer Ingelheim Investigational Site, Laval, Quebec
  - Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 2180 rue Fleury E, Montreal, Quebec
  - UHRESS, Pavillon L-C Simard, 10th Floor, Z10904, Montreal, Quebec
  - Hop du Sacre-Coeur de Montreal, Montreal, Quebec
  - Boehringer Ingelheim Investigational Site, Pointe-Claire, Quebec
  - 1401-18 Rue, Québec, Quebec
  - Boehringer Ingelheim Investigational Site, Saint-Jérôme, Quebec
  - 3001 12e ave Nord, Sherbrooke, Quebec
  - Boehringer Ingelheim Investigational Site, St-Jean Richelieu, Quebec
  - Hopital Laval, Ste-Foy, Quebec
  - Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan